CLINICAL TRIAL: NCT06138223
Title: The Effect of exeRcise And Diet on Quality of Life in Patients With Incurable Cancer of Esophagus and Stomach (RADICES)
Acronym: RADICES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Hanneke W. M. van Laarhoven, Head of Medical Oncology of Amsterdam AMC, Principal Investigator, Prof. dr. H.W.M. van Laarhoven, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL83835.018.23
Record Dates: First submitted 2023-11-02; First posted 2023-11-18 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: GastroEsophageal Cancer; Incurable Disease
Keywords: gastroesophageal cancer; GAC; Palliative; exercise intervention; nutritional intervention; Quality of life; QOL
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients randomized to the control group will receive standard medical care, including nutritional care as provided by the center in usual care. Additionally, they receive an activity tracker (like the intervention group) but without specific instructions. We will provide the control patients with written advice on physical activity and diet according to the current guidelines (in short: to avoid inactivity and be as physically active as current abilities and conditions allow, with the aim to progress towards being physically active for 150 min/week).
- Combined exercise and nutritional intervention. (Experimental): Intervention: exercise and nutrition program group
  Interventions: Other: Exercise intervention; Other: Nutrition intervention

INTERVENTIONS:
Other: Exercise intervention — During 12 weeks, patients will visit twice a week a trained oncology physiotherapist for one hour per session. This training includes supervised aerobic and resistance exercises to increase aerobic condition and muscle resistance, based on their own fitness level as assessed at baseline. Additionally, physiotherapists will educate participants on how to increase their daily activity. To this end, all participants will receive an activity tracker to monitor their daily activities.
  Arms: Combined exercise and nutritional intervention.
Other: Nutrition intervention — Once every two weeks patients in the intervention group will receive a nutritional assessment and intervention by a trained dietician for optimization of their nutritional intake to improve their nutritional status, following the ESPEN guideline on nutrition in cancer patients and the national guidelines of the National Nutritionists Oncology Working Group (NNOWG; in Dutch: Landelijke Werkgroep Diëtisten Oncologie, LWDO). Moreover, an amount of 15-25 grams of protein within 1-2 hours after exercise will be advised, to prevent muscle protein breakdown and enhance muscle protein synthesis.
  Arms: Combined exercise and nutritional intervention.

SUMMARY:
The survival of patients with incurable gastroesophageal cancer can extend over a year with anticancer therapy. However, the number of patients with deteriorating quality of life in this patient group steadily decreases over time during the treatment. Potentially reversible causes related to deterioration of quality of life are diminished muscle mass, physical capacity and nutritional status. Therefore, interventions that can target these in order to maintain or improve quality of life are urgently needed.

However, it is yet unknown whether improvement of physical capacity and nutritional status improves quality of life in patients with incurable gastroesophageal adenocarcinoma after failure of first-line treatment. Since these patients are in a precarious situation, the benefits and harms of a combined exercise and nutritional intervention should be carefully evaluated.Therefore this study investigates the effect of a combined exercise and nutrition intervention compared to usual care on quality of life in incurable GAC patients after progression upon first-line treatment.

A total of 196 patients with metastasized gastroesophageal cancer will be recruited and randomly allocated 1:1 to standard care or standard care plus a combined exercise and nutritional intervention.

DETAILED DESCRIPTION:
Randomization will be stratified based on: duration of first line therapy (shorter or longer than 6 months), WHO performance status (0, 1 versus 2), (intended) start of second-line (or further) systemic therapy for progressive disease (yes versus no) and time since failure of first line therapy (shorter or longer than 3 months ago). Due to the nature of the intervention, it is not possible to blind the patients, the local study nurses, or the investigators to the treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* Incurable adenocarcinoma of the esophagus or stomach.
* Progressive disease after first-line palliative systemic treatment OR within 6 months after completion of curative treatment (i.e. within six months after neoadjuvant chemoradiation, adjuvant nivolumab, or definitive chemoradiation for esophageal adenocarcinoma or within six months after adjuvant 5-fluorouracil, leucovorin, oxaliplatin and docetaxel (FLOT) for gastric/esophageal cancer or neoadjuvant FLOT if no adjuvant FLOT was given, or after progression during participation in the LyRICX study). Patients on capecitabine monotherapy who are eligible for oxaliplatin reintroduction can be included, too. Inclusion can take place regardless of the plan or the actual initiation of multi-line systemic treatment. (i.e. patients that have already started with second/third/etc. line therapy are eligible for inclusion too)
* Able and willing to perform the exercise and nutritional program and wear the activity tracker.
* Able and willing to fill out the POCOP/RADICES questionnaires.
* Life expectancy > 12 weeks.
* Age ≥ 18 years.

Exclusion Criteria:

* Unstable bone metastases inducing skeletal fragility as determined by the treating clinician.
* Untreated symptomatic known brain metastasis.
* Serious active infection.
* Too physically active (i.e. >210 minutes/week of moderate-to-vigorous intentional exercise) or engaging in intense exercise training comparable to the RADICES exercise program.
* Severe neurologic or cardiac impairment according to the American College of Sports Medicine criteria.
* Uncontrolled severe respiratory insufficiency as determined by the treating clinician or if the patient is dependent on oxygen suppletion in rest or during exercise.
* Uncontrolled severe pain.
* Any other contraindications for exercise as determined by the treating physician.
* Any circumstances that would impede adherence to study requirements or ability to give informed consent, as determined by the treating clinician.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life (EORTC-QLQ-30) summary score | Baseline, 6 weeks and every 12 weeks up to one year after intervention
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 item. The summary score encompasses the last question of this questionnaire.
  Scale: 1-7 Higher score means better quality of life.
  Analyzed will be the difference in quality of life between the intervention group and the control group at 12 weeks, taking into account the baseline values, and measured with the Summary Score of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30).

SECONDARY OUTCOMES:
Aerobic capacity: MSEC | Baseline, 12 weeks
  Changes in MSEC (= maximum short exercise capacity or in other words maximum wattage in the steep ramp test).
  In the steep ramp test participants cycle with a pedal frequency between 70 and 80 rpm 30 seconds at 25 W. Then every 10 seconds, the load is increased with 25 W until exhaustion. The test ends when pedal frequency falls below 60 rpm. From the MSEC peak Wattage (Wpeak) can be estimated using a regression equation.
  Scale: 0-500 W
Muscle strength: Hand grip strength | Baseline, 12 weeks
  Changes in hand grip strength. Hand grip strength: using a handgrip dynamometer the participant will be asked to squeeze the dynamometer as hard as possible for three times, for both hands. The best of three attempts for bot hands is recorded.
  Scale: 0-100 kg.
Body composition: Muscle mass | Baseline, 12 weeks
  Muscle mass will be measured with the validated InBody Dial H20B Smart Scale. Scale: 0-100 kg
Body composition: Fat mass | Baseline, 12 weeks
  Fat mass will be measured with the validated InBody Dial H20B Smart Scale. Scale: 1-100 kg
Body composition: Weight | Baseline, 12 weeks
  Weight will be measured with the validated InBody Dial H20B Smart Scale. Scale: 0-200 kg
Self-reported screening of malnutrition | Baseline and every 12 weeks up to one year after intervention
  Malnutrition will be screened using the short-form Abridged Scored Patient-Generated Subjective Global Assessment (abPG-SGA).
  Scale: 0-50 Higher score is more malnourished
Physical activity | Baseline, 12 weeks
  Physical activity is measured by an activity tracker (Fitbit). Participants are instructed to wear the tracker for 12 weeks. Mean daily steps and minutes spent in different intensity levels of physical activity are calculated, excluding no-wear days.
WHO performance status | Baseline and during the intervention, until the end of the intervention (12 weeks).
  Changes in WHO performance status.
Quality of life (EORTC-QLQ-30) total score | Baseline, 6 weeks and every 12 weeks up to one year after intervention
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 item.
  Changes in total quality of life. Scale: 0-100 Higher score means better quality of life.
Self-reported screening of sarcopenia | Baseline,12 weeks
  Changes in sarcopenia will be assessed using the Sarc-F questionnaire. (Scale 0-10, higher the score the better the condition).
Skeletal muscle index | Baseline, 12 weeks.
  Changes in skeletal muscle index, assessed by diagnostic CT-scans.
Muscle strength: leg press maximal muscle strength | Baseline, 12 weeks
  Changes in leg press one repetition maximum (1RM). Leg strength: the 12 repetition maximum is the maximum weight with which exactly 12 repetitions of a defined exercise/movement sequence can be performed with clean technique. Afterwards, the so called hypothetical 1RM (h1RM) can be calculated.
  Scale: 0-200 kg
Medical effects: Treatment toxicity | Baseline up to one year after intervention
  Changes in treatment toxicity in case of start of second line systemic treatment will be assessed using the Common Terminology Criteria for Adverse Events version 5.0
Medical effects: percentage of patients starting second-line treatment | Baseline up to one year after intervention
  Percentage of patients who have started second-line treatment
Medical effects: dose reductions | Baseline up to one year after intervention
  Treatment tolerance assessed by the amount of delivered second-line systemic treatment doses.
Medical effects: dose delays | Baseline up to one year after intervention
  Treatment tolerance assessed by the number of dose delays of second-line systemic treatment.
Medical effects: duration of systemic therapy | Baseline up to one year after intervention
  Treatment tolerance assessed by the total duration of second-line systemic treatment.
Progression-free survival | Baseline up to one year after intervention
  Time to progression
Overall survival | Baseline up to 1 year after intervention.
  Proportion of patients who have not died 1 year after baseline.
Patient reported physical activity | Baseline and every 12 weeks up to one year after intervention
  Physical activity will be assessed by the validated and reliable Short Questionnaire to assess health enhancing physical activity (SQUASH) including commuting activities, leisure time activities, household activities, and activities at work and school.
Health-related quality of life: physical functioning | Baseline and every 2 weeks during the intervention, until the end of the intervention (12 weeks).
  Changes in physical functioning, element of the EORTC-QLQ-30. To improve measurement precision compared to the standard, static EORTC-QLQ-C30 questionnaire, and to avoid floor- and ceiling effects, physical functioning will be assessed using computer adaptive testing in collaboration with experts of the EORTC.
Health-related quality of life: role functioning | Baseline and every 2 weeks during the intervention, until the end of the intervention (12 weeks).
  Changes in role functioning, element of the EORTC-QLQ-30. To improve measurement precision compared to the standard, static EORTC-QLQ-C30 questionnaire, and to avoid floor- and ceiling effects, role functioning will be assessed using computer adaptive testing in collaboration with experts of the EORTC.
Health-related quality of life: fatigue | Baseline and every 2 weeks during the intervention, until the end of the intervention (12 weeks).
  Changes in fatigue, element of the EORTC-QLQ-30. To improve measurement precision compared to the standard, static EORTC-QLQ-C30 questionnaire, and to avoid floor- and ceiling effects, fatigue will be assessed using computer adaptive testing in collaboration with experts of the EORTC.

OTHER OUTCOMES:
(Serious) Adverse Events potentially related to the exercise intervention | Baseline until the end of intervention (12 weeks)
  Adverse events will be monitored and reported according to the Exercise Harms Reporting Method (ExHaRM). Patients in both groups will be asked by the study team about adverse events systematically and in a standardized manner at the follow-up measurement. Patients will be asked by their trainer before and after each supervised session whether any (Serious) Adverse Events occurred during or since the last session (i.e. active surveillance). In addition, trainers will be asked to actively observe for adverse events that may occur during training sessions as well (i.e. passive surveillance). An adverse event panel, consisting of independent exercise and nutritional professionals and clinicians, will review all adverse event forms and determine whether adverse events are indeed potentially causally related to the exercise or nutritional intervention or not.
Adherence and compliance to the exercise and diet intervention | During the intervention period of 12 weeks
  Session attendance and adherence to the planned exercise dose/session. Deviations from the scheduled exercise dose are recorded by the physiotherapist. Attendance rates are computed as the number of supervised exercise sessions attended divided by the number of sessions prescribed and as the number of sessions with the dietician attended divided by the number of sessions prescribed. Compliance will be calculated for the exercise part as the ratio of total completed to total planned cumulative dose for three parts of the RADICES exercise program: duration of aerobic exercises, intensity of aerobic exercises and muscle strength exercises. Compliance will be calculated for the nutritional part as the ratio of total completed to total planned intake of calories, proteins and fat.
Satisfaction with the exercise and nutritional intervention | Post-intervention (12 weeks)
  Intervention group only. After the 12-week intervention period, we will assess satisfaction with the exercise and nutritional intervention by means of a self-designed questionnaire. The questionnaire contains satisfaction items with regard to the supervised exercise program, the trainer, the activity tracker and the nutritional intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke van Laarhoven, Principal Investigator — Amsterdam AMC
Locations (12):
- Netherlands (12):
  - Amsterdam UMC, Amsterdam, North Holland
  - Reinier de Graaf, Delft
  - Catharina Ziekenhuis, Eindhoven
  - Spaarne Gasthuis, Hoofddorp
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leiden Universitair Medisch Centrum, Leiden
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Laurentius Ziekenhuis, Roermond
  - Bravis Ziekenhuis, Roosendaal
  - Ikazia Ziekenhuis, Rotterdam
  - HagaZiekenhuis, The Hague
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Vulpen JK, Hiensch AE, van Hillegersberg R, Ruurda JP, Backx FJG, Nieuwenhuijzen GAP, Kouwenhoven EA, Groenendijk RPR, van der Peet DL, Hazebroek EJ, Rosman C, Wijnhoven BPL, van Berge Henegouwen MI, van Laarhoven HWM, Siersema PD, May AM. Supervised exercise after oesophageal cancer surgery: the PERFECT multicentre randomized clinical trial. Br J Surg. 2021 Jul 23;108(7):786-796. doi: 10.1093/bjs/znab078. PMID 33837380
- [Background] van Vulpen JK, Siersema PD, van Hillegersberg R, Nieuwenhuijzen GAP, Kouwenhoven EA, Groenendijk RPR, van der Peet DL, Hazebroek EJ, Rosman C, Schippers CCG, Steenhagen E, Peeters PHM, May AM. Physical ExeRcise Following Esophageal Cancer Treatment (PERFECT) study: design of a randomized controlled trial. BMC Cancer. 2017 Aug 18;17(1):552. doi: 10.1186/s12885-017-3542-8. PMID 28821284
- [Background] Hiensch AE, Monninkhof EM, Schmidt ME, Zopf EM, Bolam KA, Aaronson NK, Belloso J, Bloch W, Clauss D, Depenbusch J, Lachowicz M, Pelaez M, Rundqvist H, Senkus E, Stuiver MM, Trevaskis M, Urruticoechea A, Rosenberger F, van der Wall E, de Wit GA, Zimmer P, Wengstrom Y, Steindorf K, May AM. Design of a multinational randomized controlled trial to assess the effects of structured and individualized exercise in patients with metastatic breast cancer on fatigue and quality of life: the EFFECT study. Trials. 2022 Jul 29;23(1):610. doi: 10.1186/s13063-022-06556-7. PMID 35906659
- [Background] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Giesinger JM, Kieffer JM, Fayers PM, Groenvold M, Petersen MA, Scott NW, Sprangers MA, Velikova G, Aaronson NK; EORTC Quality of Life Group. Replication and validation of higher order models demonstrated that a summary score for the EORTC QLQ-C30 is robust. J Clin Epidemiol. 2016 Jan;69:79-88. doi: 10.1016/j.jclinepi.2015.08.007. Epub 2015 Sep 28. PMID 26327487
- [Background] Ligibel JA, Bohlke K, May AM, Clinton SK, Demark-Wahnefried W, Gilchrist SC, Irwin ML, Late M, Mansfield S, Marshall TF, Meyerhardt JA, Thomson CA, Wood WA, Alfano CM. Exercise, Diet, and Weight Management During Cancer Treatment: ASCO Guideline. J Clin Oncol. 2022 Aug 1;40(22):2491-2507. doi: 10.1200/JCO.22.00687. Epub 2022 May 16. PMID 35576506
- See also: national guidelines of the National Nutritionists Oncology Working Group (NNOWG; in Dutch: Landelijke Werkgroep Diëtisten Oncologie, LWDO) — https://nvdietist.nl/app/uploads/2021/03/Algemene_Voedings-_en_dieetbehandeling_.pdf